CLINICAL TRIAL: NCT01540461
Title: A Phase 1 Study to Determine the Safety and Pharmacokinetics of Brivanib in Chinese Subjects With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Determine the Pharmacokinetics and Safety of Brivanib in Chinese Subjects With Advanced Primary Liver Cancer (Hepatocellular Carcinoma: HCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CA182-064
Record Dates: First submitted 2012-02-23; First posted 2012-02-28 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — brivanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm: Brivanib (Experimental)
  Interventions: Drug: Brivanib

INTERVENTIONS:
Drug: Brivanib — Tablets, Oral, 800 mg, Once daily, Until withdrawal of consent, disease progression or until unmanageable toxicity
  Other Names: BMS-582664

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK), safety, and tolerability of Brivanib in Chinese subjects with Advanced Hepatocellular Carcinoma (HCC).

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

Subjects with:

* Confirmed Advanced Primary Liver Cancer (Hepatocellular Carcinoma: HCC)
* Not having received prior systemic treatment for advanced HCC
* Normal or moderately impaired liver function (Child-Pugh Class A or B (CP total score of ≤ 7))
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

Subjects with:

* Brain metastasis or evidence of leptomeningeal disease
* History of impaired brain function (encephalopathy) or active heart disease
* Unmanageable fluid in the abdomen (ascites)
* Bleeding esophageal or gastric varices within 2 months prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of Brivanib | Days 1, 2, 8, 9 and 15
Trough observed plasma concentration (Cmin) of Brivanib | Days 1, 2, 8, 9 and 15
Time of maximum observed plasma concentration (Tmax) of Brivanib | Days 1, 2, 8, 9 and 15
Area under the plasma concentration-time curve from time zero to the end of the dosing interval [AUC(TAU)] of Brivanib | Days 1, 2, 8, 9 and 15
Average steady state concentration calculated as AUC(TAU)/24 (Css_av) of Brivanib | Days 1, 2, 8, 9 and 15
Degree of fluctuation calculated as ((Cmax- Cmin)/Css_av) [Degree of fluctuation] of Brivanib | Days 1, 2, 8, 9 and 15
Terminal half-life (T-HALF) of Brivanib | Days 1, 2, 8, 9 and 15
Accumulation index calculated as the ratio: AUC(TAU) at steady-state (Day 8) divided by AUC(TAU) after the first dose (Day 1) [AI] of Brivanib | Days 1, 2, 8, 9 and 15

SECONDARY OUTCOMES:
Safety assessments based on adverse event reports and the results of vital sign measurements, electrocardiograms (ECGs), 2-D Echocardiograms, physical examinations and clinical laboratory tests | Part A: Day 1-Week 1, Day 8-Week 2, Day 15-Week 3 and Day 29-Week 5, Part B: End of treatment (approximately 24 months)
Preliminary evidence of anti-tumor activity as measured by objective response rate (ORR) and disease control rate (DCR) in Chinese subjects with advanced HCC treated with Brivanib | Screening, Week 7 and every 6 weeks up to End of treatment (approximately 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- China (3):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Harbin, Heilongjiang
  - Local Institution, Nanjing, Jiangsu

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx